CLINICAL TRIAL: NCT05455645
Title: The Therapeutic Effect of Targeted Intrinsic Foot Muscles Exercises in Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lau On Yue, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IFM exercise PF
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fasciitis, Chronic; Pain
Keywords: Strengthening; training; intrinsic foot muscle
MeSH Terms: conditions — Fasciitis, Plantar; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with one intervention arm and one control arm
Who Masked: Participant, Outcomes Assessor
Masking Description: Team members collecting outcomes data will not know participant allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted intrinsic foot muscles exercise regimen (Experimental): 4 targeted intrinsic foot exercise will be performed at least 5 times per week, once in the laboratory, and four times at home. The participants will be followed up weekly at the laboratory visit. The real-time ultrasound imaging of intrinsic foot muscles will be used as guided visual biofeedback to instruct all participants to execute all exercise movement in a correct manner. If the participant misses a session, he/she is expected to replace the lost session within the same week.
  Interventions: Other: targeted intrinsic foot muscle exercises
- Control (No Intervention): continue normal physical activity,

INTERVENTIONS:
Other: targeted intrinsic foot muscle exercises — 4 targeted intrinsic foot muscle exercises
  Arms: Targeted intrinsic foot muscles exercise regimen

SUMMARY:
A reduction of intrinsic foot muscle sizes has been identified in patients with chronic plantar fasciitis. Weaker intrinsic foot muscles has been suggested to decrease the medial longitudinal arch height and subsequently increase extra tensile stress in the plantar fascia, resulting in the chronicity of the condition. Therefore, it is speculated that atrophic intrinsic foot muscles may be a significant risk factor of developing chronic plantar fasciitis. The purpose of this study is to investigate the effect of an 8-week targeted intrinsic foot muscles exercise regimen on the intrinsic foot muscle size, symptomatic relief, and foot function improvement in long-distance runners with chronic plantar fasciitis.

DETAILED DESCRIPTION:
Distance runners are defined as running with more than 20km per week for more than 2 years. All recruited participants have > 1 year of plantar fasciitis. The diagnosis were made based on clinical symptoms and the thickness of plantar fasciitis > 4.0mm at the medial tubercle of heel by ultrasound imaging.

Arm 1: The purpose of this arm of the study is to determine if a 8-week targeted foot muscle exercise regimen, instructed with real-time ultrasound, affect the intrinsic foot muscle size, symptomatic relief, and foot function improvement of distance runners with plantar fasciitis. 32 participants will be recruited in this arm.

Arm 2: This group will not engage in any training, but will serve as a comparator for the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

1. A weekly mileage of at least 20km
2. Have running experience of at least 2 years prior to the experiment
3. if they reported tenderness on palpation of the medial calcaneal tuberosity and exhibited one of the following complaints:

   * Plantar heel pain > 1 year
   * Pain on visual analog scale of equal to or greater than 4 out of 10
   * pain on the first step in the morning or after prolonged sitting,
   * pain on prolonged standing and/or walking
   * pain when running

Exclusion Criteria:

1. Contraindications to MRI scans
2. had undergone surgery to the plantar fascia or
3. local steroid injection within the last 3 months or
4. Any of the following conditions:

   * systemic arthritis,
   * neurologic conditions
   * any coexisting painful musculoskeletal condition of the lower limb.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
muscle thickness (MT) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | baseline
  ultrasound measurement
muscle thickness (MT) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | week 4
  ultrasound measurement
muscle thickness (MT) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | week 8
  ultrasound measurement
muscle thickness (MT) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | week 12
  ultrasound measurement
cross sectional area (CSA) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | Baseline
  ultrasound measurement
cross sectional area (CSA) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | week 4
  ultrasound measurement
cross sectional area (CSA) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | week 8
  ultrasound measurement
cross sectional area (CSA) of Abductor Hallucis (AbH), Flexor hallucis brevis (FHB), Flexor digitorum brevis (FDB), quadratus plantae (QP) | week 12
  ultrasound measurement
Visual Analog Scale (VAS) pain at first steps in the morning | baseline
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) pain at first steps in the morning | week 4
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) pain at first steps in the morning | week 8
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) pain at first steps in the morning | week 12
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) worst pain of the day | baseline
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) worst pain of the day | 4
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) worst pain of the day | 8
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) worst pain of the day | 12
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Foot and Ankle Ability Measure (FAAM) | baseline
  Higher scores represent higher levels of function, with 100% representing no dysfunction.
Foot and Ankle Ability Measure (FAAM) | week 4
  Higher scores represent higher levels of function, with 100% representing no dysfunction.
Foot and Ankle Ability Measure (FAAM) | week 8
  Higher scores represent higher levels of function, with 100% representing no dysfunction.
Foot and Ankle Ability Measure (FAAM) | week 12
  Higher scores represent higher levels of function, with 100% representing no dysfunction.
Foot posture index | baseline
  Pronated postures are given a positive value, the higher the value the more pronated.
  Supinated features are given a negative value, the more negative the value the more supinated.
  For a neutral foot the final score should lie somewhere around zero
Foot posture index | week 4
  Pronated postures are given a positive value, the higher the value the more pronated.
  Supinated features are given a negative value, the more negative the value the more supinated.
  For a neutral foot the final score should lie somewhere around zero
Foot posture index | week 8
  Pronated postures are given a positive value, the higher the value the more pronated.
  Supinated features are given a negative value, the more negative the value the more supinated.
  For a neutral foot the final score should lie somewhere around zero
Foot posture index | week 12
  Pronated postures are given a positive value, the higher the value the more pronated.
  Supinated features are given a negative value, the more negative the value the more supinated.
  For a neutral foot the final score should lie somewhere around zero
Navicular Drop test | baseline
  Supinated foot (<5mm); Neutral foot (5-9mm); pronated foot (>9mm)
Navicular Drop test | week 4
  Supinated foot (<5mm); Neutral foot (5-9mm); pronated foot (>9mm)
Navicular Drop test | week 8
  Supinated foot (<5mm); Neutral foot (5-9mm); pronated foot (>9mm)
Navicular Drop test | week 12
  Supinated foot (<5mm); Neutral foot (5-9mm); pronated foot (>9mm)

SECONDARY OUTCOMES:
Postural control | baseline
  three 10-seconds eyes opened trials and three 10-seconds eyes closed trials with single-leg stance
Postural control | week 4
  three 10-seconds eyes opened trials and three 10-seconds eyes closed trials with single-leg stance
Postural control | week 8
  three 10-seconds eyes opened trials and three 10-seconds eyes closed trials with single-leg stance
Postural control | week 12
  three 10-seconds eyes opened trials and three 10-seconds eyes closed trials with single-leg stance

CONTACTS AND LOCATIONS:
Locations (1):
- CUHK-ORT Sports Injury Research Laboratory, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No